CLINICAL TRIAL: NCT06294730
Title: Coronary Microcirculation and Troponin Elevation in Septic Shock
Acronym: COMTESS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jonas Persson, Principal Investigator, Karolinska Institutet
Other Study IDs: 2018/1891-31
Record Dates: First submitted 2024-02-16; First posted 2024-03-05 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Sepsis; Myocardial Injury; Coronary Microvascular Dysfunction; Endothelial Dysfunction
Keywords: sepsis; cardiac troponin; myocardial injury; coronary microvascular dysfunction; Index of microcirculatory resistance; survival
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral plasma, serum and whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Plasma cardiac troponin (cTn) elevation is an indicator of increased mortality in patients with sepsis yet the underlying cause of troponin elevation in sepsis is not known. The COMTESS study investigates whether elevated high-sensitive cardiac Troponin T (hs-cTnT) levels in hemodynamically unstable patients with sepsis can be explained by an underlying coronary artery disease or a process within the coronary microcirculation. Fifty patients with sepsis and with hs-cTnT elevation (>15 ng/L) will undergo coronary angiography, including an assessment of coronary flow using a method called thermo-dilution to record the index of microcirculatory resistance (IMR) in the left anterior descending artery (LAD). The relationship between IMR and hs-cTnT will subsequently be analysed. It is important to identify the underlying causes of elevated cTn during sepsis to target further research with an aim to improve the survival in patients suffering from this condition.

DETAILED DESCRIPTION:
Severe sepsis and septic shock are frequent primary causes of morbidity and mortality in intensive care units worldwide with a mortality rate of 28.3 - 41.1%. Our research group has previously shown that increasing level of high-sensitive cardiac troponin T (hs-cTnT) taken in sepsis patients is associated with 30-day and one-year mortality. Importantly, our group showed that hs-cTnT is also associated with mortality during the convalescence phase (30-365-day) in sepsis survivors.

Serum cardiac troponin (cTn) measurement is used to detect myocardial injury in patients with acute ischemic heart disease. Cardiac-specific troponins (troponin I and T) are, under normal physiological conditions, only detectable in the blood in small concentrations. In the event of myocyte damage, cardiac-specific troponins I and T enter the systemic circulation and can be detected and measured using modern immunoassay methods. This has led to the use of these biomarkers to identify both the presence and even estimated extent of myocardial injury which can then in turn facilitate an early risk stratification and identification of patients suitable for coronary intervention. Since 2018, the high-sensitive cardiac troponin assays have become the recommended assays for use within the clinical setting. In stark contrast to the treatment of patients with acute myocardial infarction and elevated cTn levels, there are currently no clinical guidelines to help physicians treat, investigate or follow-up sepsis patients with sepsis-related myocardial injury.

The COMTESS study is a pioneering observational prospective clinical study of 50 critically ill sepsis patients with a sampled hs-cTnT >15 ng/L investigating the relationship between hs-cTnT level and concurrent microvascular dysfunction. Following informed consent, coronary angiography with measurements of coronary flow reserve (CFR), basal resistance index (BRI) and index of microcirculatory resistance (IMR) using thermo-dilution in the left anterior descending artery (LAD) is performed in each patient to ascertain underlying coronary microvascular dysfunction (CMVD). Fractional flow reserve (FFR) will be measured in cases where there is a coronary stenosis in the LAD. A research echocardiography is also performed on day 2-10 to examine right and left ventricular function.

Our primary hypothesis is that increasing level of hs-cTnT is associated with increasing level of CMVD in patients with sepsis and that myocardial injury thus contributes to excess death in sepsis and sepsis-survivors. The mechanisms behind myocardial injury in sepsis are not known. Disturbed sublingual microcirculatory alterations are associated with mortality in septic shock, but whether these alterations in proxy vessels translates to clinically relevant CMVD and myocardial injury in patients with sepsis is not known.

The physiological properties of endothelial cells (ECs) in the microcirculation are dependent on a complex carbohydrate-rich layer covering the EC luminal surface called the glycocalyx. Studies have shown that the disseminated dysfunctional immune response which is the hallmark of sepsis causes glycocalyx and EC injury and widespread coagulopathy leading to microvascular thrombosis. Pro-thrombotic components (e.g., neutrophile extracellular traps [NETs], and prothrombin) and components from EC and glycocalyx damage (e.g., Syndecan-1, thrombomodulin) can subsequently be analysed in plasma. Elevated level of Syndecan-1 in sepsis is associated with greater risk of death. Blood samples will be drawn during the coronary angiography for each patient and will be stored in a biobank. Our aim is to investigate if there is an association between plasma level of different microvascular components in relation to IMR level.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the Sepsis-3 definition of and diagnostic criteria for sepsis or septic shock
* Age 40 - 85 years
* Life expectancy > 1 year
* hs-cTnT values >15 ng/L

Exclusion Criteria:

* pregnancy
* previous medical history of coronary artery by-pass grafting
* heart transplant
* previously verified ejection fraction (EF) ≤39% prior to hospital admission
* Hypertrophic cardiomyopathy (Septum > 15 mm)
* severe aortic stenosis
* amyloidosis or sarcoidosis with myocardial engagement
* estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 prior to hospital admission
* asthma
* infectious endocarditis
* a medical history of abdominal, thoracic, or orthopaedic surgery within the last three months prior to hospital admission.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sepsis- or septic shock-patients with a life expectancy of >1year and non-normal high-sensitive cardiac troponin T values (>15 ng/L)
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Relationship between hs-cTnT and IMR | Day 2-10 from the onset of sepsis symptoms.
  Spline regression between the highest hs-cTnT at 0-72 hrs from vasopressor initiation and IMR at day 2-10 from sepsis onset

SECONDARY OUTCOMES:
Relationship between hs-cTnT and CFR | Day 2-10 from the onset of sepsis symptoms.
  Spline regression between the highest log hs-cTnT at 0-72 hrs from vasopressor initiation and CFR at day 2-10 from sepsis onset
Relationship between hs-cTnT and BRI | Day 2-10 from the onset of sepsis symptoms
  Spline regression between the highest hs-cTnT at 0-72 hrs from vasopressor initiation and and BRI at day 2-10 from sepsis onset
Relationship between hs-cTnT and number of diseased epicardial coronary vessels | Day 2-10 from the onset of sepsis symptoms
  ANOVA for the relationship between the highest hs-cTnT at 0-72 hrs from vasopressor initiation and number of diseased epicardial coronary vessels
Relationship between hs-cTnT and Synergy Between PCI With Taxus and Cardiac Surgery (SYNTAX)-score | Day 2-10 from the onset of sepsis symptoms
  Spline regression between the highest hs-cTnT at 0-72 hrs from vasopressor initiation and SYNTAX-score
Relationship between hs-cTnT and left ventricular end diastolic pressure (LVEDP) | Day 2-10 from the onset of sepsis symptoms
  Spline regression between the highest hs-cTnT at 0-72 hrs from vasopressor initiation and LVEDP (mmHg)
Relationship between hs-cTnT and Tricuspid annular plane systolic excursion (TAPSE) | Day 2-10 from the onset of sepsis symptoms
  Spline regression between the highest hs-cTnT at 0-72 hrs and Tricuspid annular plane systolic excursion TAPSE (mm)
Relationship between hs-cTnT and echocardiographic measurements of left ventricular global strain | Day 2-10 from the onset of sepsis symptoms
  Spline regression between the highest hs-cTnT at 0-72 hrs from vasopressor initiation and left ventricular global strain from speckle tracking (units)
Relationship between hs-cTnT and echocardiographic measurements of left diastolic dysfunction | Day 2-10 from the onset of sepsis symptoms
  ANOVA between the highest hs-cTnT at 0-72 hrs from vasopressor initiation and left ventricular diastolic function grouping (none; grade I, impaired relaxation; grade II, pseudonormalization; grade III, restrictive filling)
Relationship between measures of endothelial dysfunction and IMR | Day 2-10 from the onset of sepsis symptoms
  Spline regression between plasma levels of syndecan-1 and IMR (units)
Relationship between measures NETs and IMR | Day 2-10 from the onset of sepsis symptoms
  Spline regression between NETs in plasma and IMR

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Persson, MD, PhD, Principal Investigator — Karolinska Institutet Danderyd University Hospital
Locations (1):
- Karolinska Institutet, Danderyd University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Will be provided upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Will be provided upon reasonable request

REFERENCES:
- [Background] Lorstad S, Shekarestan S, Jernberg T, Tehrani S, Astrand P, Gille-Johnson P, Persson J. First Sampled High-Sensitive Cardiac Troponin T is Associated With One-Year Mortality in Sepsis Patients and 30- to 365-Day Mortality in Sepsis Survivors. Am J Med. 2023 Aug;136(8):814-823.e8. doi: 10.1016/j.amjmed.2023.04.029. Epub 2023 May 6. PMID 37156347
- [Background] Levy MM, Artigas A, Phillips GS, Rhodes A, Beale R, Osborn T, Vincent JL, Townsend S, Lemeshow S, Dellinger RP. Outcomes of the Surviving Sepsis Campaign in intensive care units in the USA and Europe: a prospective cohort study. Lancet Infect Dis. 2012 Dec;12(12):919-24. doi: 10.1016/S1473-3099(12)70239-6. Epub 2012 Oct 26. PMID 23103175
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Fearon WF, Nakamura M, Lee DP, Rezaee M, Vagelos RH, Hunt SA, Fitzgerald PJ, Yock PG, Yeung AC. Simultaneous assessment of fractional and coronary flow reserves in cardiac transplant recipients: Physiologic Investigation for Transplant Arteriopathy (PITA Study). Circulation. 2003 Sep 30;108(13):1605-10. doi: 10.1161/01.CIR.0000091116.84926.6F. Epub 2003 Sep 8. PMID 12963639
- [Background] De Bruyne B, Pijls NH, Smith L, Wievegg M, Heyndrickx GR. Coronary thermodilution to assess flow reserve: experimental validation. Circulation. 2001 Oct 23;104(17):2003-6. doi: 10.1161/hc4201.099223. PMID 11673336
- [Background] Fearon WF, Balsam LB, Farouque HM, Caffarelli AD, Robbins RC, Fitzgerald PJ, Yock PG, Yeung AC. Novel index for invasively assessing the coronary microcirculation. Circulation. 2003 Jul 1;107(25):3129-32. doi: 10.1161/01.CIR.0000080700.98607.D1. Epub 2003 Jun 23. PMID 12821539
- [Background] Aarnoudse W, Fearon WF, Manoharan G, Geven M, van de Vosse F, Rutten M, De Bruyne B, Pijls NH. Epicardial stenosis severity does not affect minimal microcirculatory resistance. Circulation. 2004 Oct 12;110(15):2137-42. doi: 10.1161/01.CIR.0000143893.18451.0E. Epub 2004 Oct 4. PMID 15466646
- [Background] Fearon WF, Aarnoudse W, Pijls NH, De Bruyne B, Balsam LB, Cooke DT, Robbins RC, Fitzgerald PJ, Yeung AC, Yock PG. Microvascular resistance is not influenced by epicardial coronary artery stenosis severity: experimental validation. Circulation. 2004 May 18;109(19):2269-72. doi: 10.1161/01.CIR.0000128669.99355.CB. Epub 2004 May 10. PMID 15136503
- [Background] Ong P, Camici PG, Beltrame JF, Crea F, Shimokawa H, Sechtem U, Kaski JC, Bairey Merz CN; Coronary Vasomotion Disorders International Study Group (COVADIS). International standardization of diagnostic criteria for microvascular angina. Int J Cardiol. 2018 Jan 1;250:16-20. doi: 10.1016/j.ijcard.2017.08.068. Epub 2017 Sep 8. PMID 29031990
- [Background] De Backer D, Donadello K, Sakr Y, Ospina-Tascon G, Salgado D, Scolletta S, Vincent JL. Microcirculatory alterations in patients with severe sepsis: impact of time of assessment and relationship with outcome. Crit Care Med. 2013 Mar;41(3):791-9. doi: 10.1097/CCM.0b013e3182742e8b. PMID 23318492
- [Background] Fernandez-Sarmiento J, Molina CF, Salazar-Pelaez LM, Florez S, Alarcon-Forero LC, Sarta M, Hernandez-Sarmiento R, Villar JC. Biomarkers of Glycocalyx Injury and Endothelial Activation are Associated with Clinical Outcomes in Patients with Sepsis: A Systematic Review and Meta-Analysis. J Intensive Care Med. 2023 Jan;38(1):95-105. doi: 10.1177/08850666221109186. Epub 2022 Jun 19. PMID 35722738
- [Background] Piotti A, Novelli D, Meessen JMTA, Ferlicca D, Coppolecchia S, Marino A, Salati G, Savioli M, Grasselli G, Bellani G, Pesenti A, Masson S, Caironi P, Gattinoni L, Gobbi M, Fracasso C, Latini R; ALBIOS Investigators. Endothelial damage in septic shock patients as evidenced by circulating syndecan-1, sphingosine-1-phosphate and soluble VE-cadherin: a substudy of ALBIOS. Crit Care. 2021 Mar 19;25(1):113. doi: 10.1186/s13054-021-03545-1. PMID 33741039
- [Background] Sun T, Wang Y, Wu X, Cai Y, Zhai T, Zhan Q. Prognostic Value of Syndecan-1 in the Prediction of Sepsis-Related Complications and Mortality: A Meta-Analysis. Front Public Health. 2022 Apr 11;10:870065. doi: 10.3389/fpubh.2022.870065. eCollection 2022. PMID 35480580
- [Background] Colicchia M, Perrella G, Gant P, Rayes J. Novel mechanisms of thrombo-inflammation during infection: spotlight on neutrophil extracellular trap-mediated platelet activation. Res Pract Thromb Haemost. 2023 Mar 11;7(2):100116. doi: 10.1016/j.rpth.2023.100116. eCollection 2023 Feb. PMID 37063765
- [Background] Cox D. Sepsis - it is all about the platelets. Front Immunol. 2023 Jun 7;14:1210219. doi: 10.3389/fimmu.2023.1210219. eCollection 2023. PMID 37350961